CLINICAL TRIAL: NCT02294032
Title: The Role of B Cells in Kidney Allograft Dysfunction
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5140147; GCAT 2014 (Other Grant/Funding Number: GCAT 2014)
Record Dates: First submitted 2014-05-29; First posted 2014-11-19 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Kidney; Complications, Allograft; Transplantation Infection
Keywords: Bcells; kidney allograft dysfunction; antibody mediated rejection
MeSH Terms: interventions — Immunosuppressive Agents; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, and plasma or serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney Transplant: Patients who are about to undergo a kidney transplant and are on immunosuppressive agents.
  Interventions: Drug: Immunosuppressive Agents

INTERVENTIONS:
Drug: Immunosuppressive Agents — standard of care for patients post-transplant
  Other Names: Prograf, Cellcept

SUMMARY:
The purpose of this study is to understand the role of specific B cells in activating or repressing an anti-allograft immune response after kidney transplantation. In this study, blood will be collected from kidney transplant patients during different timepoints, prior to and after their transplant. Knowledge gained from study findings will be used to develop therapeutic strategies to prevent antibody-mediated rejection, which is a major cause of long-term graft loss in kidney transplant patients.

DETAILED DESCRIPTION:
The purpose of this study is to understand the role of specific B cells in activating or repressing an anti-allograft immune responses after kidney transplantation. This study aims to address two major challenges in kidney transplantation: 1. to guide physicians when immunosuppressive drugs are weaned, and 2. to identify patients who are at risk or in the process of developing antibody-mediated rejection. In this study, blood will be collected from kidney transplant patients during different timepoints, prior to and after their transplant. Knowledge gained from study findings will be used to develop therapeutic strategies to prevent antibody-mediated rejection, which is a major cause of long-term graft loss in kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign the written informed consent form (ICF). For pediatric patients, a parent or legal guardian must sign ICF
* Either a Kidney or Liver transplant patient: 1) on the waitlist or 2) transplanted
* Healthy volunteer samples collected to use as the control group for statistical validity

Exclusion Criteria:

* Inability to make all of the required long-term post-transplant visits.
* Females who are pregnant or nursing a child
* Liver patients with hepatitis C virus

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and Adult patients who are on the waitlist for a kidney or liver, or are about to undergo kidney or liver transplantation.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Blood collection prior to and after kidney transplantation | 1,3,6,12,18,24,36,48, and 60 months
  Blood will be collected from kidney transplant patients prior to and after their transplant (1-, 3-, 6-, 12-, 18-, 24-, 36-, 48-, and 60- months post-transplant). We will try to better understand the role of specific B-cells after kidney transplant by using enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
B cell count | Up to 60 months
  For each patient, we will be measuring the frequency of cells from each B cell subset within the total peripheral blood mononuclear cells (PBMNCs) by MACSQuant cell counts. The distribution of B cells subsets within the total B cell pool will also be determined. Mean Fluorescence Intensity (MFI) of activation markers (CD86 and CD69) on B cells will also be compared across the samples.

CONTACTS AND LOCATIONS:
Overall Officials: Michael de Vera, MD, FACS, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Transplantation Institute, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seron D, Moreso F, Arias M, Campistol JM, Curto J, Hernandez D, Morales JM, Sanchez-Fructuoso A, Abraira V; Spanish Late Allograft Dysfunction Study Group. Estimation of renal allograft half-life: fact or fiction? Nephrol Dial Transplant. 2011 Sep;26(9):3013-8. doi: 10.1093/ndt/gfq788. Epub 2011 Feb 3. PMID 21292814
- [Background] Colvin RB, Hirohashi T, Farris AB, Minnei F, Collins AB, Smith RN. Emerging role of B cells in chronic allograft dysfunction. Kidney Int Suppl. 2010 Dec;(119):S13-7. doi: 10.1038/ki.2010.436. PMID 21116310
- [Background] Newell KA, Asare A, Kirk AD, Gisler TD, Bourcier K, Suthanthiran M, Burlingham WJ, Marks WH, Sanz I, Lechler RI, Hernandez-Fuentes MP, Turka LA, Seyfert-Margolis VL; Immune Tolerance Network ST507 Study Group. Identification of a B cell signature associated with renal transplant tolerance in humans. J Clin Invest. 2010 Jun;120(6):1836-47. doi: 10.1172/JCI39933. Epub 2010 May 24. PMID 20501946
- [Background] Sagoo P, Perucha E, Sawitzki B, Tomiuk S, Stephens DA, Miqueu P, Chapman S, Craciun L, Sergeant R, Brouard S, Rovis F, Jimenez E, Ballow A, Giral M, Rebollo-Mesa I, Le Moine A, Braudeau C, Hilton R, Gerstmayer B, Bourcier K, Sharif A, Krajewska M, Lord GM, Roberts I, Goldman M, Wood KJ, Newell K, Seyfert-Margolis V, Warrens AN, Janssen U, Volk HD, Soulillou JP, Hernandez-Fuentes MP, Lechler RI. Development of a cross-platform biomarker signature to detect renal transplant tolerance in humans. J Clin Invest. 2010 Jun;120(6):1848-61. doi: 10.1172/JCI39922. Epub 2010 May 24. PMID 20501943
- [Background] Halloran PF. Immunosuppressive drugs for kidney transplantation. N Engl J Med. 2004 Dec 23;351(26):2715-29. doi: 10.1056/NEJMra033540. No abstract available. PMID 15616206
- [Background] Barnett AN, Hadjianastassiou VG, Mamode N. Rituximab in renal transplantation. Transpl Int. 2013 Jun;26(6):563-75. doi: 10.1111/tri.12072. Epub 2013 Feb 18. PMID 23414100
- [Background] Rehnberg M, Amu S, Tarkowski A, Bokarewa MI, Brisslert M. Short- and long-term effects of anti-CD20 treatment on B cell ontogeny in bone marrow of patients with rheumatoid arthritis. Arthritis Res Ther. 2009;11(4):R123. doi: 10.1186/ar2789. Epub 2009 Aug 17. PMID 19686595
- [Background] Everly MJ. Understanding and addressing the humoral immune response in transplant recipients. Clin Transpl. 2012:225-7. No abstract available. PMID 23721026
- [Background] Everly MJ. Immunosuppression regimens to address alloantibodies in transplant recipients. Clin Transpl. 2012:219-23. PMID 23721025
- [Background] Kannabhiran D, Everly MJ, Walker-McDermott JK, Tiongko S, Friedlander R, Putheti P, Sharma V, Dadhania D. Changes in IgG subclasses of donor specific anti-HLA antibodies following bortezomib-based therapy for antibody mediated rejection. Clin Transpl. 2012:229-35. PMID 23721027
- [Background] Thibault-Espitia A, Foucher Y, Danger R, Migone T, Pallier A, Castagnet S, G-Gueguen C, Devys A, C-Gautier A, Giral M, Soulillou JP, Brouard S. BAFF and BAFF-R levels are associated with risk of long-term kidney graft dysfunction and development of donor-specific antibodies. Am J Transplant. 2012 Oct;12(10):2754-62. doi: 10.1111/j.1600-6143.2012.04194.x. Epub 2012 Aug 6. PMID 22883025
- [Background] Xu H, He X, Liu Q, Chen Y, Zhu Y, Shi D, Zhang X. The abnormal high expression of B cell activating factor belonging to TNF superfamily (BAFF) and its potential role in kidney transplant recipients. Cell Mol Immunol. 2008 Dec;5(6):465-70. doi: 10.1038/cmi.2008.58. PMID 19118513
- [Background] Clatworthy MR, Espeli M, Torpey N, Smith KG. The generation and maintenance of serum alloantibody. Curr Opin Immunol. 2010 Oct;22(5):669-81. doi: 10.1016/j.coi.2010.08.018. PMID 20932734
- [Background] Stegall MD, Raghavaiah S, Gloor JM. The (re)emergence of B cells in organ transplantation. Curr Opin Organ Transplant. 2010 Aug;15(4):451-5. doi: 10.1097/MOT.0b013e32833b9c11. PMID 20613525
- [Background] Lynch RJ, Silva IA, Chen BJ, Punch JD, Cascalho M, Platt JL. Cryptic B cell response to renal transplantation. Am J Transplant. 2013 Jul;13(7):1713-23. doi: 10.1111/ajt.12308. Epub 2013 Jun 10. PMID 23750851
- [Background] Anolik JH, Looney RJ, Lund FE, Randall TD, Sanz I. Insights into the heterogeneity of human B cells: diverse functions, roles in autoimmunity, and use as therapeutic targets. Immunol Res. 2009 Dec;45(2-3):144-58. doi: 10.1007/s12026-009-8096-7. Epub 2009 Apr 7. PMID 19350211
- [Background] Kaminski DA, Wei C, Qian Y, Rosenberg AF, Sanz I. Advances in human B cell phenotypic profiling. Front Immunol. 2012 Oct 10;3:302. doi: 10.3389/fimmu.2012.00302. eCollection 2012. PMID 23087687
- [Background] Anolik JH, Barnard J, Cappione A, Pugh-Bernard AE, Felgar RE, Looney RJ, Sanz I. Rituximab improves peripheral B cell abnormalities in human systemic lupus erythematosus. Arthritis Rheum. 2004 Nov;50(11):3580-90. doi: 10.1002/art.20592. PMID 15529346
- [Background] Iwata S, Saito K, Tokunaga M, Yamaoka K, Nawata M, Yukawa S, Hanami K, Fukuyo S, Miyagawa I, Kubo S, Tanaka Y. Phenotypic changes of lymphocytes in patients with systemic lupus erythematosus who are in longterm remission after B cell depletion therapy with rituximab. J Rheumatol. 2011 Apr;38(4):633-41. doi: 10.3899/jrheum.100729. Epub 2010 Dec 15. PMID 21159836
- [Background] Kinnunen T, Chamberlain N, Morbach H, Cantaert T, Lynch M, Preston-Hurlburt P, Herold KC, Hafler DA, O'Connor KC, Meffre E. Specific peripheral B cell tolerance defects in patients with multiple sclerosis. J Clin Invest. 2013 Jun;123(6):2737-41. doi: 10.1172/JCI68775. Epub 2013 May 15. PMID 23676463
- [Background] Sanz I, Wei C, Lee FE, Anolik J. Phenotypic and functional heterogeneity of human memory B cells. Semin Immunol. 2008 Feb;20(1):67-82. doi: 10.1016/j.smim.2007.12.006. Epub 2008 Feb 6. PMID 18258454
- [Background] Moens L, Wuyts M, Meyts I, De Boeck K, Bossuyt X. Human memory B lymphocyte subsets fulfill distinct roles in the anti-polysaccharide and anti-protein immune response. J Immunol. 2008 Oct 15;181(8):5306-12. doi: 10.4049/jimmunol.181.8.5306. PMID 18832686
- [Background] Gambichler T, Tigges C, Burkert B, Hoxtermann S, Altmeyer P, Kreuter A. Absolute count of T and B lymphocyte subsets is decreased in systemic sclerosis. Eur J Med Res. 2010 Jan 29;15(1):44-6. doi: 10.1186/2047-783x-15-1-44. PMID 20159671
- [Background] Adams AB, Newell KA. B cells in clinical transplantation tolerance. Semin Immunol. 2012 Apr;24(2):92-5. doi: 10.1016/j.smim.2011.08.019. Epub 2011 Sep 29. PMID 21958959
- [Background] Bloom D, Chang Z, Pauly K, Kwun J, Fechner J, Hayes C, Samaniego M, Knechtle S. BAFF is increased in renal transplant patients following treatment with alemtuzumab. Am J Transplant. 2009 Aug;9(8):1835-45. doi: 10.1111/j.1600-6143.2009.02710.x. Epub 2009 Jun 12. PMID 19522878
- [Background] Shlipak MG, Matsushita K, Arnlov J, Inker LA, Katz R, Polkinghorne KR, Rothenbacher D, Sarnak MJ, Astor BC, Coresh J, Levey AS, Gansevoort RT; CKD Prognosis Consortium. Cystatin C versus creatinine in determining risk based on kidney function. N Engl J Med. 2013 Sep 5;369(10):932-43. doi: 10.1056/NEJMoa1214234. PMID 24004120
- [Background] Iwata Y, Matsushita T, Horikawa M, Dilillo DJ, Yanaba K, Venturi GM, Szabolcs PM, Bernstein SH, Magro CM, Williams AD, Hall RP, St Clair EW, Tedder TF. Characterization of a rare IL-10-competent B-cell subset in humans that parallels mouse regulatory B10 cells. Blood. 2011 Jan 13;117(2):530-41. doi: 10.1182/blood-2010-07-294249. Epub 2010 Oct 20. PMID 20962324
- [Background] Lehnhardt A, Dunst F, van Husen M, Loos S, Oh J, Eiermann T, Koch M, Kemper MJ. Elevated serum levels of B-cell activating factor in pediatric renal transplant patients. Pediatr Nephrol. 2012 Aug;27(8):1389-95. doi: 10.1007/s00467-012-2142-8. Epub 2012 Mar 28. PMID 22453734
- [Background] Banham G, Prezzi D, Harford S, Taylor CJ, Hamer R, Higgins R, Bradley JA, Clatworthy MR. Elevated pretransplantation soluble BAFF is associated with an increased risk of acute antibody-mediated rejection. Transplantation. 2013 Aug 27;96(4):413-20. doi: 10.1097/TP.0b013e318298dd65. PMID 23842189
- [Background] Thien M, Phan TG, Gardam S, Amesbury M, Basten A, Mackay F, Brink R. Excess BAFF rescues self-reactive B cells from peripheral deletion and allows them to enter forbidden follicular and marginal zone niches. Immunity. 2004 Jun;20(6):785-98. doi: 10.1016/j.immuni.2004.05.010. PMID 15189742
- [Background] Woodland RT, Schmidt MR. Homeostatic proliferation of B cells. Semin Immunol. 2005 Jun;17(3):209-17. doi: 10.1016/j.smim.2005.02.006. PMID 15826826
- [Background] Smith SH, Cancro MP. Cutting edge: B cell receptor signals regulate BLyS receptor levels in mature B cells and their immediate progenitors. J Immunol. 2003 Jun 15;170(12):5820-3. doi: 10.4049/jimmunol.170.12.5820. PMID 12794106
- [Background] Kandala NB, Connock M, Grove A, Sutcliffe P, Mohiuddin S, Hartley L, Court R, Cummins E, Gordon C, Clarke A. Belimumab: a technological advance for systemic lupus erythematosus patients? Report of a systematic review and meta-analysis. BMJ Open. 2013 Jul 19;3(7):e002852. doi: 10.1136/bmjopen-2013-002852. Print 2013. PMID 23872289
- [Background] Vadasz Z, Toubi E. [Belimumab--the biological drug for systemic lupus erythematosus: as discussed during the American College of Rheumatology (ACR) conference - 2012]. Harefuah. 2013 May;152(5):304-6. No abstract available. Hebrew. PMID 23885457